CLINICAL TRIAL: NCT03698812
Title: A Multicenter Prospective Follow-up Study on the Effect of Histological Remission on the Clinical Prognosis of Ulcerative Colitis
Brief Title: A Multicenter Prospective Cohort Study on the Clinical Prognosis of Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xinying wang, vice-professor, Nanfang Hospital, Southern Medical University
Other Study IDs: LC2016PY007
Record Dates: First submitted 2018-09-30; First posted 2018-10-09 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Prospective Study; Ulcerative Colitis in Remission
Keywords: Ulcerative Colitis; Mucosal Healing; Histological Remission; Prospective Study
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Colonoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen retention will be kept as evidence to evaluate the condition of health.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- CTL group: control group
  Interventions: Combination Product: Colonoscope
- EXP group: Colonoscope
  Interventions: Combination Product: Colonoscope

INTERVENTIONS:
Combination Product: Colonoscope — take off specimen

SUMMARY:
Mucosal healing or histological remission is an important target for the treatment of inflammatory bowel disease. In this study, patients with mucosal healing are defined as a control group, observing their clinical outcomes for 3 years, and describing the recurrence rate. The secondary objective is to study the operative rate, glucocorticoid utilization rate, treatment escalation rate, hospitalization rate and incidence of related complications.

DETAILED DESCRIPTION:
Assess the health condition of patients for 1year, 2year,3year and analyze outcomes and complications.

ELIGIBILITY:
Inclusion Criteria:

* sign informed consent before proceeding with any specific procedure.
* ages:14-75
* subjects were diagnosed with ulcerative colitis in written form. (written diagnosis should include at least one histopathological change).
* mucosal healing or histological remission has been achieved after medical treatment.

  1. histological assessment is performed by 2 pathologists independently, and endoscopy have been independently evaluated by two endoscopic doctors.
  2. prospective cohort study (3) definition of endoscopic mucosal healing: Baron score<=1 and Mayo score<=1 (4) definition of histological remission: Truelove/ Richards=1 and Geboes score<3.0 (5) sampling methods: the terminal ileum, the ascending colon, the transverse colon, the descending colon, the sigmoid colon, and the rectum, the six parts were randomly taken specimen (at least 2 tissues each).
* data integrity: the research data include: 1) enteroscopy; 2) laboratory examination indicators: blood routine, erythrocyte sedimentation rate, C reaction protein, liver function, renal function, fecal calprotectin, 3) serum concentration of infliximab, antibody to infliximab.
* subjects were treated with the following treatment Mesalazine, glucocorticoid, immunosuppressive agent (azathioprine or thalidomide), biologics (infliximab) 7. subjects have the ability to answer the questionnaire

Exclusion Criteria:

* The diagnosis is unclear
* Subjects with history of colectomy
* Subjects with history of cancerogenesis
* Subjects with severe liver disease, defined as child-pugh Grade B or Grade C
* Subjects with severe renal disease, defined as Estimated glomerular filtration rate<30
* major cardiovascular events, such as stroke, myocardial infarction, or unstable angina, occurred within 3 months before enrollment.
* Subjects during pregnancy.
* alcohol or drug abuse
* poor compliance 10 Planners and investors

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The project includes 320 cases from 4 Hospital. The EG and CG
  has 160 cases. Nanfang Hospital of southern medical university:230 cases(EG115,CG115) Zhujiang Hospital of southern medical university:30 cases(EG15,CG15) Third affiliated hospital of southern medical university： 30 cases(EG15,CG15) First Hospital Affiliated to Shantou University：30 cases(EG15,CG15)
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
relapse rate | 1year
  CAI ≥5 or necessity for additional treatment

SECONDARY OUTCOMES:
surgery rate | 1year，2year，3year
  disease progress requiring surgery
Rehospitalization rate | 1year，2year，3year
  observation
requirement for escalation of drugs | 1year，2year，3year
  observation
complication rate | 1year，2year，3year
  toxic megacolon，perforation，carcinogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
1. ages:14-75
  2. subjects were diagnosed with ulcerative colitis in written form. (written diagnosis should include at least one histopathological change).
  3. mucosal healing or histological remission has been achieved after medical treatment.
  4. data integrity
Supporting Information: Study Protocol
Time Frame: 1year,2year,3year
Access Criteria: patients with ulcerative colitis in histological remission.

REFERENCES:
- [Result] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735